CLINICAL TRIAL: NCT05368909
Title: Assessment of the Effects of a Dietary Supplement on the Sleep Health and Sleep Quality of People With Sleep Problems: A Randomized, Double-blind, Placebo-controlled, Crossover Design Study
Brief Title: Clinical Study to Assess a Dietary Supplement on Sleep Health and Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 4Life Research, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 4Life-Sleep
Record Dates: First submitted 2022-05-02; First posted 2022-05-10 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Sleep Quality; Sleep Health
Keywords: Sleep Health; Sleep Quality; Melatonin; Lavender essential oil; GABA
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 before Cross Over (Experimental): Participants were randomized and divided into two groups: Supplement Group and Placebo Group. In this Arm 1, participants first go through a 1-week washout period, and then take either Supplement or Placebo as assigned for 2 week.
  Interventions: Dietary Supplement: Sleep Supplement; Dietary Supplement: Placebo
- Arm 2 after Cross Over (Experimental): In Arm 2, Supplement Group and Placebo Group cross over. After a 1-week washout period, and both group will take whatever product they did not take in Arm 2, for 2 week.
  Interventions: Dietary Supplement: Sleep Supplement; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Sleep Supplement — Proprietary sleep formula containing Tri Factor, Ashwagandha root extract, Lavender, Pyridoxal-5-Phosphate, Melatonin, gamma aminobutyric acid (GABA) and Magnesium.
Dietary Supplement: Placebo — Placebo product

SUMMARY:
The primary objective of this study is to evaluate the effects of a proprietary oral supplement on the sleep health and quality of people with sleep problems. It is a double-blinded placebo-controlled crossover clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers
* Judged by the Investigator to be in general good health on the basis of medical history
* Willing to wash out of all dietary supplements, essential oils, and non-prescription sleep aids or Rx sleep aids for the duration of the study
* Insomnia Severity Index score of ≥ 8
* Must agree to maintain the same eating, exercise, and sleep arrangements for the whole duration of the study

Exclusion Criteria:

* Pregnant and/or lactating women
* Known allergy or adverse reaction to ingredients in the product: Tri Factor (bovine colostrum and egg yolk extracts), Ashwagandha root extract, Lavender, Pyridoxal-5-Phosphate, Melatonin, gamma aminobutyric acid (GABA) or Magnesium
* Prescription sedative or psychoactive (including anti-depressant) medication use
* Diagnosis of a sleep disorder (e.g., sleep apnea, periodic limb movement disorder, etc.) or high clinical probability of another sleep disorder based on sleep history
* A clinically unstable medical condition as defined by a new diagnosis or change in medical management in the previous 4 months (e.g., myocardial infarction, congestive heart failure, Cheyne-Stokes breathing, unstable angina, thyroid disease, depression or psychosis, ventricular arrhythmias, cirrhosis, surgery, or recently diagnosed cancer)
* Routine consumption of more than 2 alcoholic beverages per day or consumption of caffeine past 2 PM for the duration of the study
* Illicit drug use
* Use of prescription stimulants (modafinil, dextroamphetamine, etc.)
* Use of prescription medications known to affect sleep (antidepressants, anti-anxiety, opioids, alpha-blockers, beta-blockers, corticosteroids, ACE inhibitors, angiotensin II-receptor blockers, cholinesterase inhibitors, allergy medication, asthma medication, glucosamine and chondroitin, statins, anti-smoking or thyroid medication, muscle relaxants, anticonvulsants)
* Unable to perform tests due to inability to communicate verbally, inability to write and read in English; less than a 10th grade reading level; visual, hearing or upper extremity motor deficit
* Night shift workers in situations or occupations where they regularly experience jet lag, or have irregular work schedules by history over the last 6 months
* Unwilling to consume or unable to swallow capsules/tablets
* Previous exposure to this product in earlier testing phases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Saliva Melatonin level changes | 6 weeks
  Samples taken before bedtime at night and 2 hours after wakeup the next morning. A total of 8 samples were taken for each subject: (2) right after first washout, (2) right after Arm 1, (2) right after the second washout, (2) right after Arm 2.
Insomnia Severity Index Score | 6 weeks
  A scale used to measure the severity of insomnia. Total score categories:
  0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)

SECONDARY OUTCOMES:
Sleep Onset Latency | 6 weeks
  Sleep latency, or sleep onset latency, is the time it takes a person to fall asleep after turning the lights out.
Total Sleep Time | 6 weeks
  Total time a person spends asleep over a given night
Sleep Efficiency | 6 weeks
  Sleep efficiency is typically referring to the percentage of time a person spends asleep at night. To calculate this, you take a ratio of the total amount of time a person was asleep on a given night divided by the total amount of time they spent in bed, then multiply that by 100 to create a percentage.
Leeds Sleep Evaluation Questionnaire (LSEQ) Score | 6 weeks
  A 10-item, subjective, self-report measure, the LSEQ was designed to assess changes in sleep quality over the course of a psychopharmacological treatment intervention. The scale evaluates four domains: ease of initiating sleep, quality of sleep, ease of waking, and behavior following wakefulness. Total LSEQ Score ranges from 0 to 100, with 100 being the worst sleep quality and health overall.

CONTACTS AND LOCATIONS:
Locations (1):
- 4Life Research, Sandy City, Utah, United States

IPD SHARING:
Plan to Share IPD: No